CLINICAL TRIAL: NCT00182156
Title: Cohort Study Examining the Effects of Short Daily Hemodialysis As Compared to Conventional Hemodialysis in Outpatients Treated at St Joseph's Healthcare, Hamilton
Brief Title: Cohort Study Comparing Short Daily Hemodialysis (HD) With Conventional HD
Status: Withdrawn | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Azim Gangji, Associate professor, McMaster University
Other Study IDs: Nephrology Divisional Funds
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: End-stage Renal Disease; Thrombocytopathy; Cardiovascular Diseases
Keywords: hemodialysis; platelet function analyzer; bioimpedance; pulse wave velocity; end stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic; Blood Platelet Disorders; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: conventional HD
- 2: short daily HD
- 3: PD

SUMMARY:
This study is examining the effects of short daily hemodialysis on platelet function, fluid volume control, arterial stiffness and patient quality of life, as compared to conventional hemodialysis.

DETAILED DESCRIPTION:
Bleeding is a common cause of morbidity and mortality in patients with end stage renal disease. A major cause of uremic bleeding is due to platelet dysfunction. It has been theorized that in renal failure, toxins accumulate, some of which inhibit primary hemostasis. All aspects of normal platelet function are affected. Platelet function has previously been difficult to quantify but recently a novel test, the platelet function analyzer (PFA-100) has been determined to be both sensitive and specific in assessing platelet function. Conventional hemodialysis (CHD) has been shown to partially correct thrombocytopathy. Enhanced uremic clearance can now be attained through the use of short daily hemodialysis (SDHD). Cardiovascular disease is the most common cause of mortality in dialysis patients, accounting for 40% of deaths. Volume overload is associated with high blood pressure, left ventricular hypertrophy and elevated markers of inflammation and these factors have been associated with increased cardiovascular mortality. SDHD has been shown to control blood pressure and limit volume expansion. Pulse wave velocity (PWV) has been used to assess arterial compliance and reduction of arterial elasticity of large and small arteries which have been associated with cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient is enrolled in short daily hemodialysis program
* Patient is minimum of 18 years old

Exclusion Criteria:

* Patient is unable to consent due to language barrier
* Patient is unable to consent due to cognitive difficulties
* Patient refuses consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Short daily HD v PD v conventional HD
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-10; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Azim Gangji, MD, Principal Investigator — Clinical Scholar, Medicine; Catherine M Clase, MD, Principal Investigator — Associate Professor, Medicine
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada